CLINICAL TRIAL: NCT04535011
Title: PRACT: A Pragmatic Randomized Adaptive Clinical Trial to Investigate Controlling Alcohol Related Harms in a Low-Income Setting; Emergency Department Brief Interventions in Tanzania
Brief Title: PRACT to Investigate Controlling Alcohol Related Harms in a Low-Income Setting; Emergency Department BIs in Tanzania
Acronym: PRACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00103724; R01AA027512 (NIH)
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Use Disorder; Injury Traumatic; Trauma
MeSH Terms: conditions — Alcoholism; Wounds and Injuries | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Study Phase 1: The investigators will evaluate whether PPKAY with personalized text booster or PPKAY with standard text booster will reduce the quantity or frequency of alcohol use, the number of binge drinking events or the number of alcohol-related consequences based on the Drinker Inventory of Consequences (DrInC) compared to usual care.
  Study Phase 2: The investigators will evaluate whether PPKAY alone is an inferior supplement to PPKAY plus standard or personalized text booster
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care (No Intervention): No prevention or educational information verbally or written coinciding with current usual care
- PPKAY (Experimental): One-time, 15-minute, nurse-led motivational interview discussing safe drinking behaviors, and negotiating change in alcohol use
  Interventions: Behavioral: PPKAY (brief intervention)
- PPKAY with Standard Booster (Experimental): One-time, 15-minute, nurse-led motivational interview discussing safe drinking behaviors, and negotiating change in alcohol use.
  Weekly standard text booster until final follow-up (e.g., "Reducing your alcohol intake to less than 4 drinks per day reduces your risk of alcohol-related consequences")
  Interventions: Behavioral: PPKAY (brief intervention); Behavioral: Standard Booster
- PPKAY with Personalized Booster (Experimental): One-time, 15-minute, nurse-led motivational interview discussing safe drinking behaviors, and negotiating change in alcohol use Weekly personalized text booster until final follow-up (e.g., "Remember to reduce your alcohol less than 4 drinks to achieve your goal of… [being a better husband].")
  Interventions: Behavioral: PPKAY (brief intervention); Behavioral: Personalized Booster

INTERVENTIONS:
Behavioral: PPKAY (brief intervention) — PPKAY is a nurse-administered, one-on-one, 15-minute brief intervention (BI) for alcohol use using FRAMES motivational interviewing techniques. The BI is a four-step discussion: 1) Raise the Subject of Alcohol, 2) Provide Feedback, 3) Enhance Motivation 4) Negotiate and Advice.
  Arms: PPKAY; PPKAY with Personalized Booster; PPKAY with Standard Booster
Behavioral: Standard Booster — After discharge from the hospital, a standard motivational text message will be sent to their cell phone twice monthly for the duration of the study. In a rotating fashion, one of four standard motivational texts translated into Swahili will be sent to their cell phones.
  Arms: PPKAY with Standard Booster
Behavioral: Personalized Booster — After discharge from the hospital, a personalized motivational text message will be sent to participant cell phones twice monthly for the duration of the study. In a rotating fashion, one of four personalized motivational texts will be sent to their cell phones. Personalized texts will be created with the content obtained from the motivational interview sessions. At each session, the research nurse conducting the intervention will record four messages based on the content of the session to be sent as the Personalized Booster.
  Arms: PPKAY with Personalized Booster

SUMMARY:
Alcohol use is rapidly increasing in low- and middle-income countries, where it is inexpensive, readily available, poorly regulated, and there are few resources devoted to promoting safe alcohol use. A Brief Intervention based on a motivational interviewing framework has been shown to reduce alcohol use and alcohol-related harms. The investigators have translated and adapted a Brief Intervention for alcohol to the Tanzanian context and Swahili language called "Punguza Pombe Kwa Afya Yako (PPKAY)/ Reduce Alcohol for Your Health." This project will evaluate this intervention in injury patients presenting for care at the Kilimanjaro Christian Medical Center in Moshi, Tanzania. By using innovative adaptive clinical trial methods, the investigators will expedite the development of the most effective way to integrate this intervention into clinical care. By the end of this project, investigators will have identified the most effective brief intervention components and be able to characterize the intervention's effect overall. Additionally, investigators will standardize adaptive trial methods to revolutionize the science of clinical trials for behavioral sciences in low-resource settings.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age)
* present seeking initial care at the KCMC ED for an acute (<24 hours) injury
* not clinically intoxicated (i.e., have capacity to consent).
* one or more of the following: 1) disclosed alcohol use prior to injury, 2) scored ≥8 on the AUDIT, 3) test positive (>0.0 g/dL) by alcohol breathalyzer.

Exclusion Criteria:

* do not speak the native Swahili language
* too ill or unable to communicate
* prior enrollment in this study
* decline informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in number of binge drinking days (previous 4 weeks) | Baseline, 3 months, 6 months, 9 months, 12 months, 24 months

SECONDARY OUTCOMES:
Change in frequency of alcohol use (previous 2 weeks) | Baseline, 3 months, 6 months, 9 months, 12 months, 24 months
Change in quantity of alcohol use (previous 2 weeks) | Baseline, 3 months, 6 months, 9 months, 12 months, 24 months
Change in alcohol-related harms measured by the Drinker Inventory of Consequences (DrInC) | Baseline, 3 months, 6 months, 9 months, 12 months, 24 months
  The Drinker Inventory of Consequences (DrInC) is a fifty-item questionnaire with scores ranging from 0 to 150, where a higher number indicates a greater number of negative consequences.
Change in alcohol use disorder | Baseline, 3 months, 6 months, 9 months, 12 months, 24 months
  Alcohol use disorder measured with AUDIT (alcohol use disorder identification test) score. AUDIT is a ten-item tool, with scores ranging from 0 to 40, where a higher score indicates higher risk alcohol use.
Change in depression | Baseline, 3 months, 6 months, 9 months, 12 months, 24 months
  Depression measured with Patient Health Questionnaire 9 (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Staton, MD, Principal Investigator — Duke University
Locations (1):
- Kilimanjaro Christian Medical Centre, Moshi, Kilimanjaro, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staton CA, Minja L, de Souza JVP, Gallis JA, Santos PCP, Buono M, Sakita F, Ngowi K, Boshe J, Phillips AJ, Vissoci JRN, Mmbaga BT. Effectiveness of a brief intervention and text-based booster in the emergency department to reduce harmful and hazardous alcohol use: A pragmatic randomized adaptive clinical trial in Moshi, Tanzania. PLoS Med. 2025 Oct 27;22(10):e1004548. doi: 10.1371/journal.pmed.1004548. eCollection 2025 Oct. PMID 41144564
- [Derived] Staton CA, Agnihotri D, Phillips AJ, Ngowi K, Huo L, Boshe J, Sakita F, Tupetz A, Suffoletto B, Mmbaga BT, Vissoci JRN. Development of culturally-appropriate text message booster content to follow a brief intervention focused on reducing alcohol related harms for injury patients in Moshi, Tanzania. PLOS Glob Public Health. 2024 Jul 25;4(7):e0002717. doi: 10.1371/journal.pgph.0002717. eCollection 2024. PMID 39052647
- [Derived] Staton CA, Zadey S, O'Leary P, Phillips A, Minja L, Swahn MH, Hirshon JM, Boshe J, Sakita F, Vissoci JRN, Mmbaga BT. PRACT: a pragmatic randomized adaptive clinical trial protocol to investigate a culturally adapted brief negotiational intervention for alcohol use in the emergency department in Tanzania. Trials. 2022 Feb 5;23(1):120. doi: 10.1186/s13063-022-06060-y. PMID 35123566

DOCUMENTS (1):
  • Informed Consent Form (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT04535011/ICF_001.pdf